CLINICAL TRIAL: NCT00055549
Title: The Effects of an NMDA-Receptor Antagonist in Idiopathic Voice Disorders
Brief Title: Dextromethorphan to Treat Patients With Voice Spasms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030119; 03-N-0119
Record Dates: First submitted 2003-03-05; First posted 2003-03-05 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-11-13

CONDITIONS: Voice Disorders
Keywords: Dextromethorphan; Sensorimotor Modulation; Spasmodic Dysphonia; Muscular Tension Dysphonia; Voice Tremor; Lorazepam; Dysphonia; Macular Tension Dysphonia
MeSH Terms: conditions — Voice Disorders; Dysphonia | interventions — Dextromethorphan; Lorazepam

INTERVENTIONS:
Drug: Dextromethorphan
Drug: Lorazepam

SUMMARY:
This study will examine how dextromethorphan, a drug that alters reflexes of the larynx (voice box), might change voice symptoms in people with voice disorders due to uncontrolled laryngeal muscle spasms. These include abductor spasmodic dysphonia (breathy voice breaks), adductor spasmodic dysphonia (vowel breaks), muscular tension dysphonia (tight strained voice), and vocal tremor (tremulous voice). Dextromethorphan-one of a group of drugs called NMDA antagonists-has been used for years in over-the-counter cough suppressant medicines. In animal studies, the drug has blocked one of the reflexes in the larynx that may be associated with spasms in the laryngeal muscles. This study will compare the effects of dextromethorphan, lorazepam (a valium-type drug), and a placebo (inactive substance) in patients with the four types of voice disorders described above.

Patients with spasmodic dysphonia, muscular tension dysphonia and vocal tremor may be eligible for this study. Individuals who smoke or use tobacco, who have vocal nodules or polyps, or who have a history of airway obstruction may not participate. Candidates will be screened with a medical history and physical examination, a questionnaire, voice recording (repeating sentences into a microphone), and nasolaryngoscopy (examination of the larynx with a tube advanced through the nose). For the nasolaryngoscopy, the inside of the nose is sprayed with a decongestant (to open the nasal passages) and possibly a local anesthetic. A small, flexible tube called a nasolaryngoscope is passed through the nose to look at the larynx during speech and other tasks, such as singing, whistling and prolonged vowels.

Participants will be admitted to the NIH Clinical Center for each of three visits, which will last from the afternoon of one day to late afternoon of the following day. At each visit, patients will complete a questionnaire, baseline speech recording, and a test for sedation level. They will take three pills-either dextromethorphan, lorazepam, or placebo-one every 6 hours. Vital signs will be checked every 6 hours and the level of sedation during waking hours will be monitored. One to three hours after taking the third pill, speech recording, questionnaire and test of sedation will be repeated to check for possible voice changes. Patients will be given a different pill at each visit.

...

DETAILED DESCRIPTION:
Studies of spasmodic dysphonia (SD) have increasingly pointed to the possibility of a central sensori-motor control disorder. Sensori-motor processing has been found abnormal in both adductor and abductor spasmodic dysphonia based on reflex conditioning studies. These studies demonstrated an increased frequency of R2 muscle responses during rapid paired presentation of electrical stimuli to the superior laryngeal nerve in spasmodic dysphonia. Thus, uncontrolled R2 responses were hypothesized to be the basis for the uncontrolled muscle bursts in these patients. Selective suppression of late R2 laryngeal adductor responses by N-methyl-D-Aspartate (NMDA) blockade in cats was demonstrated by Ambalavanar et.al. In particular, dextromethorphan reduced the frequency of R2 responses from 95% to 25% (P = 0.015). Dextromethorphan is a widely used antitussive agent that has been in use for over 30 years. In a double-blind randomized crossover design, 3 groups of patients will receive be randomly assigned to one of 6 order cohorts. They will then receive either dextromethorphan at a 8 mg/kg/d dose divided in a Q6 hour dosing schedule with only 3 doses administered PO every 6 hours for 3 dosages, 04 mg/kg/d of lorazepam PO every 6 hours for 3 dosages or a placebo administrated in the same way during Phase A. After a minimum of a 1-week washout interval, the patients will be given either the other medication or placebo during Phase B and then the remaining medication or placebo during Phase C.

Our hypothesis is that dextromethorphan, an NMDA receptor blocker, will reduce voice breaks in spasmodic dysphonia to a greater degree than lorazepam, which has similar sedating side effects, but does not affect NMDA receptors with a different mechanism. On the other hand, patients with other idiopathic voice disorders, muscular tension dysphonia and vocal tremor, are hypothesized not to have a similar benefit from dextromethorphan. During the double-blind randomized cross-over study, three groups will be included, 10 patients with adductor or abductor spasmodic dysphonia, 10 with muscular tension dysphonia and 10 with vocal tremor. The results will determine if dextromethorphan has potential as a treatment option for patients with adductor or abductor SD.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with Spasmodic Dysphonia will meet the following criteria:

1. No structural abnormalities affecting the larynx such as vocal fold nodules, polyps, carcinoma, cysts, contact ulcers, inflammation (laryngitis).
2. Symptoms of adductor or abductor spasmodic dysphonia present during speech and not apparent at rest,
3. Symptoms of adductor or abductor spasmodic dysphonia less evident during whisper, singing or falsetto.
4. Symptoms of adductor or abductor spasmodic dysphonia become worse with prolonged speaking, practice or anxiety.
5. Reflexive and emotional aspects of voice function are unaffected, such as coughing and laughter or crying.

Patients with Muscular Tension Dysphonia will meet the following criteria:

1. Increased phonatory muscle tension in the paralaryngeal and suprahyoid muscles on palpation,
2. Constant elevation of the larynx in the neck during speech.
3. A consistent hypertonic laryngeal posture for phonation, either an open posterior glottic chink between the arytenoid cartilages on phonation, an anterior-posterior squeeze (pin hole posture) or ventricular hyperadduction.
4. A normally appearing larynx.

Patients with vocal tremor will have tremor isolated to the larynx without noticeable tremor of the head and pharynx. Tremor of the vocal folds should be evident during a prolonged vowel and also noticeable in the larynx during connected speech containing vowels.

EXCLUSION CRITERIA:

Subjects in all three groups will be without:

1. Cardiac, pulmonary, neurological, psychiatric or speech and hearing problems as determined by medical history and examination by a physician and an EKG. Any patient with a history of airway obstruction will be excluded from the study.
2. Reduction in the range of vocal fold movement during non-speech tasks such as whistling suggesting either paralysis or paresis, joint abnormality or neoplasm.
3. No smokers or tobacco users will be included in the study.
4. Exclude mucosal changes such as vocal nodules or polyps.
5. Subjects with a history of a psychiatric disorder, under the care of a psychiatrist, or on medications for treatment of a psychiatric disorder will be excluded from study. Examples of psychiatric disorders to be excluded are: somatoform disorders, conversion disorders, currently under treatment for a major depression, or a history of schizophrenia or a bipolar disorder. However, a history of a previous episode of a minor reactive depression would not exclude a person from participation.
6. Subjects taking carbonic anhydrase inhibitors, cimetidine, hydrochlorthiazide, nicotine, quinidine, ranitidine, sodium or calcium bicarbonate and triamterene must either discontinue these medications or be excluded from study.
7. Subjects with grade 2 or higher hepatic or renal dysfunction will be excluded from study.
8. Pregnant women will be excluded from the study as it is not known if the study drugs are harmful to the fetus. If a woman becomes pregnant during the study, she will be removed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65
Dates: Start 2003-03-04; Primary Completion 2009-11-13 (Actual); Study Completion 2009-11-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ambalavanar R, Ludlow CL, Wenthold RJ, Tanaka Y, Damirjian M, Petralia RS. Glutamate receptor subunits in the nucleus of the tractus solitarius and other regions of the medulla oblongata in the cat. J Comp Neurol. 1998 Dec 7;402(1):75-92. PMID 9831047
- [Background] Ambalavanar R, Purcell L, Miranda M, Evans F, Ludlow CL. Selective suppression of late laryngeal adductor responses by N-methyl-D-aspartate receptor blockade in the cat. J Neurophysiol. 2002 Mar;87(3):1252-62. doi: 10.1152/jn.00595.2001. PMID 11877499
- [Background] Aminoff MJ, Dedo HH, Izdebski K. Clinical aspects of spasmodic dysphonia. J Neurol Neurosurg Psychiatry. 1978 Apr;41(4):361-5. doi: 10.1136/jnnp.41.4.361. PMID 650244